CLINICAL TRIAL: NCT01989546
Title: Pilot Trial of BMN 673, an Oral PARP Inhibitor, in Patients With Advanced Solid Tumors and Deleterious BRCA Mutations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alice Chen, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140015; 14-C-0015
Record Dates: First submitted 2013-11-16; First posted 2013-11-21 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Advanced Ovarian Cancer; Primary Peritoneal Cancer; Advanced Breast Cancer; Advanced Solid Tumors
Keywords: DNA Damage; Advanced Solid Tumors; BRCA Mutations; PARP Inhibitor; Pharmacodynamics
MeSH Terms: interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Talazoparib (BMN 673) (Experimental): Single agent
  Interventions: Drug: BMN 673

INTERVENTIONS:
Drug: BMN 673 — Poly (ADP-ribose) polymerase (PARP) inhibitor; has been shown to cause single-agent synthetic lethality in breast cancer 1 and breast cancer 2 (BRCA1/2)- and phosphatase and tensin homolog (PTEN)-deficient cell lines, and has potent antitumor activity in animal models of tumors harboring mutations in deoxyribonucleic acid (DNA) repair pathways.
  Other Names: Talazoparib

SUMMARY:
Background:

* The poly (ADP-ribose) polymerase (PARP) family of enzymes is critical for maintaining genomic stability by regulating a variety of deoxyribonucleic acid (DNA) damage repair mechanisms.
* Talazoparib (BMN 673) is a PARP inhibitor with greater in vitro activity than any other PARP inhibitor currently in development. BMN 673 has been shown to cause single-agent synthetic lethality in breast cancer 1 and breast cancer 2 (BRCA1/2)- and phosphatase and tensin homolog (PTEN)-deficient cell lines and has potent antitumor activity in animal models of tumors harboring mutations in DNA repair pathways.
* BMN 673 is showing promising single-agent activity in patients with advanced ovarian and breast cancer harboring deleterious BRCA mutations.
* This pilot study will evaluate the pharmacodynamic effects of BMN 673 on DNA damage and apoptosis markers in tumor biopsy tissue.

Primary Objective:

-Determine the pharmacodynamic effect of BMN 673 in tumor biopsies from patients with advanced ovarian, breast, or other solid tumor and deleterious BRCA mutations.

Secondary Objectives:

* Determine the response rate (Complete Response (CR) + Partial Response (PR) of treatment with BMN 673 in patients with advanced ovarian or primary peritoneal carcinoma and deleterious BRCA mutations.
* Determine the response rate (CR + PR) of treatment with BMN 673 in patients with advanced breast carcinoma and deleterious BRCA mutations.
* Determine the response rate (CR + PR) of treatment with BMN 673 in patients with advanced solid tumor (other than breast or ovarian) and deleterious BRCA mutations.

Eligibility:

* Adult patients with documented deleterious BRCA 1 or 2 mutations with histologically confirmed ovarian, primary peritoneal, breast, prostate, pancreas, gastric or other solid tumor whose disease has progressed following at least one standard therapy or who have no acceptable standard treatment options.
* No major surgery, radiation, or chemotherapy within 4 weeks prior to study enrollment, and recovered from toxicities of prior therapies to at least eligibility levels.
* Age greater than or equal to 18 years of age; Eastern Cooperative Oncology Group (ECOG) performance status less than equal to 2
* Adequate organ function.
* Willingness to undergo tumor biopsies.

Study Design:

* BMN 673 will be administered orally each day in 28-day cycles.
* Dosing will be at the established recommended Phase II dose of 1000 mcg/day each day for

  28 days.
* We plan to accrue a total of 12 evaluable patients per cohort for a total of 36 patients. To allow for some patients who will not be evaluable, the accrual ceiling is 42 patients.
* Tumor biopsies will be mandatory at baseline (pre-dose), and then approximately 3-6 hours post BMN 673 on day 8. An optional tumor biopsy may also be collected at time of disease progression.

SCHEMA

* BMN 673 is administered orally each day in 28-day cycles
* Tumor biopsies will be performed at baseline (pre-treatment) and 3-6 hrs post dose on cycle 1 day 8. An optional tumor biopsy may also be collected at time of disease progression. Tumor biopsies will be evaluated for protease activated receptor (PAR) levels, DNA damage response markers such as >=H2A.X Variant Histone (H2AX), cleaved caspase 3, excision repair cross-complementing group 1 (ERCC1), pNbs1, XPF, RAD51, and pT1989ATR, and, as indicators of ataxia telangiectasia and Rad3-related protein (ATR)/ataxia telangiectasia mutated (ATM) activation, Checkpoint kinase 1 (chk1) and Checkpoint kinase 2 (chk2)
* Blood samples for circulating tumor cells (CTC) analyses will be collected at baseline (pre-treatment), on cycle 1 day 1(3-6 hours post dose), on cycle 1 day 8 (3-6 hours post dose), and on cycle 2 day 1 (3-6 hours post dose)
* Blood samples for pharmacokinetic (PK) analysis will be collected on cycle 1 day 1 pre-dose and 0.5, 1, 2, 3, 4, 6,8, and 24 hours post-dose, on cycle 1 day 8 (3-6 hours post dose), and on cycle 2 day 1 pre-dose and 3-6 hours post dose.

DETAILED DESCRIPTION:
Background:

* The poly (ADP-ribose) polymerase (PARP) family of enzymes is critical for maintaining genomic stability by regulating a variety of deoxyribonucleic acid (DNA) damage repair mechanisms.
* Talazoparib (BMN 673) is a PARP inhibitor with greater in vitro activity than any other PARP inhibitor currently in development. Talazoparib (BMN 673) has been shown to cause single-agent synthetic lethality in breast cancer 1 and breast cancer 2 (BRCA1/2)- and phosphatase and tensin homolog (PTEN)-deficient cell lines, and has potent antitumor activity in animal models of tumors harboring mutations in DNA repair pathways.
* Talazoparib (BMN 673) is showing promising single-agent activity in patients with advanced ovarian and breast cancer harboring deleterious BRCA mutations.
* This pilot study will evaluate the pharmacodynamic effects of talazoparib (BMN 673) on DNA damage and apoptosis markers in tumor biopsy tissue.

Primary Objective:

-Determine the pharmacodynamic effect of talazoparib (BMN 673) in tumor biopsies from patients with advanced ovarian, breast, or other solid tumor and deleterious BRCA mutations.

Secondary Objectives:

-Determine the response rate (Complete Response (CR) + Partial Response (PR) of treatment with talazoparib (BMN 673) in patients with deleterious BRCA mutations.

Eligibility:

* Adult patients with documented deleterious BRCA 1 or 2 mutations with histologically confirmed ovarian, primary peritoneal, breast, prostate, pancreas, gastric or other solid tumor whose disease has progressed following at least one standard therapy or who have no acceptable standard treatment options.
* No major surgery, radiation, or chemotherapy within 4 weeks prior to study enrollment, and recovered from toxicities of prior therapies to at least eligibility levels.
* Age greater than or equal to 18 years of age; Eastern Cooperative Oncology Group (ECOG) performance status less than equal to 2
* Adequate organ function.
* Willingness to undergo tumor biopsies.

Study Design:

* Talazoparib (BMN 673) will be administered orally each day in 28-day cycles.
* Dosing will be at the established recommended Phase II dose of 1000 microgram/day each day for 28 days.
* To meet the primary, pharmacodynamic endpoint of the trial, we plan to accrue a total of 12 patients with matched, evaluable baseline and day 8 biopsies. To allow for some patients whose biopsies will not be evaluable (i.e., will contain <5% tumor content), the accrual ceiling is 24 patients. The number of patients evaluable for objective response, while relevant to the secondary objective of the trial, will not be considered in determining completion of accrual.
* Tumor biopsies will be mandatory at baseline (pre-dose), and then approximately 3-6 hours post talazoparib (BMN 673) on day 8. One optional tumor biopsy may also be collected either on day 1 (+/- 2 days) of the cycle following any restaging at which a 10-19% increase in tumor volume is observed (according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria) if the patient has been on study for at least 4 cycles, or at time of disease progression.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adult patients with documented deleterious breast cancer 1 and breast cancer 2 (BRCA 1 or 2) mutations with histologically confirmed ovarian, primary peritoneal, breast, prostate, pancreas, gastric or other solid tumor whose disease has progressed following at least one standard therapy or who have no acceptable standard treatment options.

Patients with ovarian cancer should have one prior platinum-based

chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound. This initial treatment may have included intraperitoneal therapy, consolidation, biologic/targeted (noncytotoxic) agents or extended therapy administered after surgical or non-surgical

assessment. Ovarian cancer patients with both platinum-sensitive and platinum resistant disease are eligible. Patients with platinum-refractory disease are NOT eligible.

Patients with metastatic disease must have received at least one line of standard of care (SOC) treatment for metastatic disease prior to enrollment

* Age greater than or equal to 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin less than or equal to 1.5 times institutional upper limit of normal
  * Aspartate aminotransferase (AST) Serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) Serum glutamic pyruvic transaminase (SGPT) less than or equal to 3 times institutional upper limit of normal
  * creatinine less than or equal to 1.5 times institutional upper limit of normal

OR

--creatinine clearance greater than or equal to 60 mL/min for patients with creatinine levels above institutional normal.

The effects of BMN 673 on the developing human fetus are unknown. For this reason and because PARP inhibitors are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days after completing study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 3 months after completion of BMN 673 administration.

* Patients must be able to swallow whole tablets or capsules. Nasogastric or G-tube administration is not allowed. Any gastrointestinal disease which would impair ability to swallow, retain, or absorb drug is not allowed.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients with human epidermal growth factor receptor 2 (HER2)-positive advanced breast cancer or ovarian cancer should have received at least two lines of systemic therapy in the advanced setting.
* Patients with prostate cancer can continue to receive treatment with Gonadotropin-releasing hormone (GnRH) agonists while on study, as long as there is evidence of disease progression on therapy.

EXCLUSION CRITERIA:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Patients who have had prior treatment with any PARP inhibitors are ineligible.
* Patients who are receiving any other investigational agents.
* Patients with known active brain metastases or carcinomatous meningitis are excluded from this clinical trial. Patients whose brain metastatic disease status has remained stable for greater than or equal to 4 weeks following treatment of brain metastases are eligible to participate at the discretion of the principal investigator.
* Eligibility of subjects receiving any medications or substances with the potential to affect the activity or pharmacokinetics of BMN 673 will be determined following review by the principal investigator.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the effects of the study drugs on the developing fetus are unknown.
* human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with BMN 673. In addition, these patients are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients who require use of coumarin-derivative anticoagulants such as warfarin are excluded. Low molecular weight heparin is permitted for prophylactic or therapeutic use. Low-dose warfarin (less than or equal to 1 mg/day) is permitted.
* Women who are currently lactating

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Litton JK, Rugo HS, Ettl J, Hurvitz SA, Goncalves A, Lee KH, Fehrenbacher L, Yerushalmi R, Mina LA, Martin M, Roche H, Im YH, Quek RGW, Markova D, Tudor IC, Hannah AL, Eiermann W, Blum JL. Talazoparib in Patients with Advanced Breast Cancer and a Germline BRCA Mutation. N Engl J Med. 2018 Aug 23;379(8):753-763. doi: 10.1056/NEJMoa1802905. Epub 2018 Aug 15. PMID 30110579
- [Background] de Bono J, Ramanathan RK, Mina L, Chugh R, Glaspy J, Rafii S, Kaye S, Sachdev J, Heymach J, Smith DC, Henshaw JW, Herriott A, Patterson M, Curtin NJ, Byers LA, Wainberg ZA. Phase I, Dose-Escalation, Two-Part Trial of the PARP Inhibitor Talazoparib in Patients with Advanced Germline BRCA1/2 Mutations and Selected Sporadic Cancers. Cancer Discov. 2017 Jun;7(6):620-629. doi: 10.1158/2159-8290.CD-16-1250. Epub 2017 Feb 27. PMID 28242752
- [Result] Wilsker DF, Barrett AM, Dull AB, Lawrence SM, Hollingshead MG, Chen A, Kummar S, Parchment RE, Doroshow JH, Kinders RJ. Evaluation of Pharmacodynamic Responses to Cancer Therapeutic Agents Using DNA Damage Markers. Clin Cancer Res. 2019 May 15;25(10):3084-3095. doi: 10.1158/1078-0432.CCR-18-2523. Epub 2019 Feb 21. PMID 30792217
- [Derived] Mittra A, Coyne GHOS, Zlott J, Kummar S, Meehan R, Rubinstein L, Juwara L, Wilsker D, Ji J, Miller B, Navas T, Ferry-Galow KV, Voth AR, Chang TC, Jiwani S, Parchment RE, Doroshow JH, Chen AP. Pharmacodynamic effects of the PARP inhibitor talazoparib (MDV3800, BMN 673) in patients with BRCA-mutated advanced solid tumors. Cancer Chemother Pharmacol. 2024 Mar;93(3):177-189. doi: 10.1007/s00280-023-04600-0. Epub 2023 Nov 27. PMID 38010394
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0015.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Talazoparib (BMN 673): Single-agent BMN 673 (talazoparib) dosed orally at 1 mg/day in 28-day cycles. This poly (ADP-ribose) polymerase (PARP) inhibitor has been shown to cause single-agent synthetic lethality in breast cancer 1 and breast cancer 2 (BRCA1/2)- and phosphatase and tensin homolog (PTEN)-deficient cell lines, and has potent antitumor activity in animal models of tumors harboring mutations in deoxyribonucleic acid (DNA) repair pathways.
Period: Overall Study
Arm/Group | Talazoparib (BMN 673)
Started | 9
Completed | 0
Not Completed | 9
Not completed — Clinical Progression | 1
Not completed — Disease progression on study | 8

BASELINE CHARACTERISTICS:
Arm/Group | Talazoparib (BMN 673)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.23 (12.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Achieve a Sustained Progressive Disease (PD) Response, Defined to be at Least 4% Nuclear Area Positive (NAP) γH2AX at the Day 8 Biopsy
Description: Evaluation of drug effect on deoxyribonuclecic acid (DNA) damage response will be performed using immunofluorescence assays to measure the DNA damage repair marker γH2A (the phosphorylated form of histone family member X, H2AX) in the nucleus of tumor cells obtained via core biopsy.
Time Frame: Cycle 1, day 8
Measure: Number; unit: percentage of participants
Arm/Group | Talazoparib (BMN 673)
Number analyzed (Participants) | 9
percentage of participants | 44.4

2. Secondary Outcome: Response Rate (Complete Response (CR) + Partial Response (PR) of Treatment With Talazoparib (BMN 673) in Participants With Deleterious Breast Cancer (BRCA) Mutations
Description: Response will be evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST)1. 1 guidelines; restaging scans will be carried out every 2 cycles. Complete Response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. And progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: Restaging scans will be carried out every 2 cycles (8 weeks) until the end of treatment (average, 7 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib (BMN 673)
Number analyzed (Participants) | 9
Participants
  Complete Response | 0
  Partial Response | 5

3. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 28 months and 24 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib (BMN 673)
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 28 months and 24 days.
Arm/Group | Talazoparib (BMN 673)
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Talazoparib (BMN 673) (N=9)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Talazoparib (BMN 673) (N=9)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Activated partial thromboplastin time prolonged (Investigations) | 4 (5)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 2 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 6 (33)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Bloating (Gastrointestinal disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (11)
Dizziness (Nervous system disorders) | 3 (8)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Edema limbs (General disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Eye disorders - Other, Eye disorder; let eye itching (Eye disorders) | 1 (1)
Fatigue (General disorders) | 4 (5)
Fever (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 2 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (4)
Hot flashes (Vascular disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 8 (32)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (10)
Neutrophil count decreased (Investigations) | 6 (22)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 2 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Palpitations (Cardiac disorders) | 2 (2)
Platelet count decreased (Investigations) | 8 (19)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Renal calculi (Renal and urinary disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical and medical procedures - Other, Surgical and medical procedure - Bronchoscopy (Surgical and medical procedures) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5)
Weight loss (Investigations) | 3 (5)
White blood cell decreased (Investigations) | 8 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT01989546/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT01989546/ICF_001.pdf